CLINICAL TRIAL: NCT03103672
Title: Comparison of Inhalation Anesthesia and Total Intravenous Anesthesia in Percutaneous Transhepatic Cholangiography
Brief Title: Total Intravenous Anesthesia in Percutaneous Transhepatic Cholangiography
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Yusuf Ziya ÇOLAK, Department of Anesthesiology, Inonu Univercity, School of Medicine, Inonu University
Other Study IDs: 2016/101
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Percutaneous Transhepatic Cholangiography
Keywords: quality of anesthesia; reduce recovery time

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Groupe I: Patients who will receive inhalation anesthesia
  Interventions: Procedure: Percutaneous transhepatic cholangiography
- Groupe 2: Patients who will receive total intravenous anesthesia
  Interventions: Procedure: Percutaneous transhepatic cholangiography

INTERVENTIONS:
Procedure: Percutaneous transhepatic cholangiography — Percutaneous transhepatic cholangiography (PTC) can be performed via the right midaxillary approach, though a subxiphoid approach is occasionally needed
  Other Names: PTC

SUMMARY:
Percutaneous transhepatic cholangiography is a disturbing procedure for patients.

TIVA with short-acting anesthetics such as propofol and remifentanil is characterized by hemodynamic stability and better compilation profile The purpose of this study; To compare total intravenous anesthesia with inhalation anesthesia in patients undergoing percutaneous transhepatic cholangiography under general anesthesia.

DETAILED DESCRIPTION:
Percutaneous transhepatic cholangiography is a disturbing procedure for patients. Especially pain at the time of dilation can be a serious problem. These situations may be required local anesthetics, intravenous narcotics and sedatives or general anesthesia (1).

TIVA with short-acting anesthetics such as propofol and remifentanil is characterized by hemodynamic stability and better compilation profile (2).

The purpose of this study; To compare total intravenous anesthesia with inhalation anesthesia in patients undergoing percutaneous transhepatic cholangiography under general anesthesia and Determine their advantages and disadvantages.

1. Michael J. Lee, Peter R. Mueller, Sanjay Saini, Peter F. Hahn, Stewen L. Dawson. Percutaneous Dilatation of Benign Biliary Strictures: Single-Season Therapy with General Anesthesia. AJR: 157, December 1991: 1263-1266
2. Xiaoqian Deng, Tao Zhu. Clinical comparison of propofol-remifentanil TCI with sevoflurane induction / maintenance anesthesia in laparoscopic cholecystectomy. Pak J Med Sci 2014 Vol. 30 No. 5: 1017-1021

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing percutaneous transhepatic cholangiography with general anesthesia

Exclusion Criteria:

* Essential data were missing
* Patient participating in other research projects
* Drug allergy
* Anesthetic complication story

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing percutaneous transhepatic cholangiography
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01-02 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Recovery time from anesthesia | up to postoperative 1 hours
  Time for Modified Aldrete Score 9 and over

SECONDARY OUTCOMES:
Heart rate | up to postoperative 1 hours
  Every 5 minutes during the process
Mean blood pressure | up to postoperative 1 hours
  Every 5 minutes during the process

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Z Çolak, MD, Principal Investigator — Department of Anesthesia, İnonu Univercity, School of Medicine

IPD SHARING:
Plan to Share IPD: No